CLINICAL TRIAL: NCT03215927
Title: A Randomized, Controlled Pilot Trial to Evaluate the Efficacy and Safety of Subcutaneous Abatacept in Treating Interstitial Lung Disease Associated With the Anti-synthetase Syndrome
Brief Title: Abatacept for the Treatment of Myositis-associated Interstitial Lung Disease
Acronym: ATtackMy-ILD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rohit Aggarwal, MD (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Rohit Aggarwal, MD, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY19030443; BMS: IM101-657 (Other Grant/Funding Number: BMS)
Record Dates: First submitted 2017-06-28; First posted 2017-07-12 (Actual); Results first posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Myositis; Interstitial Lung Disease
Keywords: ILD
MeSH Terms: conditions — Myositis; Lung Diseases, Interstitial | interventions — Abatacept

STUDY DESIGN:
Intervention Model Description: A 1:1 randomization scheme for abatacept 125 mg vs. placebo as a weekly subcutaneous (SQ) injection for 24 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only the site pharmacist is unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Placebo Comparator): Subcutaneous placebo injection weekly for 24 weeks.
  Interventions: Other: Placebo
- Abatacept (Experimental): Subcutaneous injection of abatacept 125 mg weekly for 24 weeks. 24 week optional follow up phase all subjects receive abatacept 125 mg weekly.
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — Abatacept 125mg subcutaneous weekly
  Other Names: Orencia
  Arms: Abatacept
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
A randomized, controlled pilot trial to evaluate the efficacy and safety of subcutaneous Abatacept in treating interstitial lung disease associated with the anti-synthetase syndrome.

DETAILED DESCRIPTION:
This is a proof of concept study to evaluate the efficacy, safety and tolerability of abatacept in Syn-ILD in a multi-center randomized, placebo-controlled 6-month (24-week) pilot study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Anti-synthetase syndrome defined as the patient possessing 1 antisynthetase autoantibody (Jo-1, PL-12, PL-7, KS, OJ, EJ, Zo) in the presence of autoimmune ILD.
3. ILD defined by radiographic (HRCT chest) findings of reticulation, honeycombing or ground glass opacities (GGO) without another plausible explanation. HRCT chest defining ILD for inclusion criteria, should be within last 1 year done as SOC.
4. Active ILD (see Section 4.2).
5. Baseline FVC a) % <80% b) FVC 80-100% with > = 10% decline in FVC in last 12 months as minimal threshold of ILD severity (PFT done within last 3 months is acceptable for inclusion criteria determination)
6. SOC immunosuppressive therapy (IS) therapy:

   1. Steroids (prednisone or other forms of steroid in equivalent doses) OR one of the other immunosuppressive agent (either Mycophenolate (MMF) or Azathioprine (AZA) OR a combination of steroid and an immunosuppressive agent. MMF (maximum of 3 gm/day) or azathioprine (maximum of 200 mg/day).Goal is to start the trial drug (or placebo) soon after starting SOC (MMF/AZA/Steroids) and their doses are stable. Note that patients on steroids alone as well as not on steroids can be enrolled in the trial as well.
   2. Desired dose of the SOC therapy should be reached 4 weeks prior to first study visit (Visit 1). No dose changes are allowed 4 weeks prior to first study visit.
   3. Dose of concomitant therapy (SOC) cannot be changed during the 24 weeks of the trial unless safety/toxicity issues supervene.
   4. If on steroid, the steroid dose must be stable for 2 weeks prior to Visit 1.
7. No other concomitant IS medications including methotrexate, cyclosporine, intravenous immunoglobulin (IVIG), tacrolimus, cyclophosphamide or tofacitinib.
8. No concomitant biologic agents (i.e. rituximab, anti-tumor necrosis factor (TNF) agents, tocilizumab).
9. Additional IS therapy: Patient cannot begin any new IS therapy or new steroid taper for the 24-week study period, except if severe clinical worsening (flare up) of the disease requiring rescue therapy occurs (i.e. documentation of worsening of PFT/HRCT and patient and physician determination of worsening). See section of rescue medication below for details.
10. If the enrolling physician is planning to discontinue current IS agent or steroid before clinical trial, then following washout period is required prior to Visit 1.

    Medication Washout Period methotrexate 4 weeks Other IS agent (e.g. azathioprine, cyclosporine, tacrolimus, leflunomide, mycophenolate mofetil) 4 weeks IVIg or cyclophosphamide 3 months rituximab 6 months infliximab or adalimumab 8 weeks glucocorticoids 2 weeks etanercept 2 weeks anakinra 1 week pirfenidone 4 weeks
11. Men and women of reproductive potential must agree to use an acceptable method of birth control during the trial period.
12. Subject has provided written informed consent.

Exclusion Criteria:

A patient will be excluded if any of the following Exclusion Criteria are met:

1. Severe end stage lung disease:

   1. FVC ≤30% or Forced expiratory volume (FEV1) ≤ 30% or
   2. Requirement of high O2 requirement ≥ 6 L/min at rest for >1 month before the study enrollment or
   3. Listed for lung transplantation or
   4. PI feels that ILD is severe and end stage fibrosis is such that there is low potential for improvement with any disease modifying intervention.
2. Subjects under the age of 18.
3. Known active current or history of recurrent bacterial, viral, fungal, mycobacterial or other infections (including but not limited to tuberculosis and atypical mycobacterial disease, hepatitis B and C, and herpes zoster, but excluding fungal infections of nail beds).
4. Any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening.
5. Active tuberculosis (TB) requiring treatment within the previous 3 years. Patients should be screened for latent TB using purified protein derivative (PPD)/or quantiferon gold within last 1 year and, if positive, treated following local practice guidelines prior to initiating abatacept (ABT). Patients treated for active tuberculosis with no recurrence in 3 years are permitted.
6. Primary or secondary immunodeficiency (history of or currently active) unless related to primary disease under investigation.
7. Pregnant women or nursing (breast feeding) mothers.
8. History of alcohol, drug or chemical abuse within 1 year prior to screening or any medical condition or physical or psychological state that the PI feels would not allow the subject to safely complete the study.
9. Major surgery (including joint surgery) within 8 weeks prior to screening or planned major surgery within 6 months following randomization.
10. Treatment with any other investigational agent within 4 weeks (or 5 half-lives of the investigational drug, whichever is longer) of screening.
11. Previous treatment with the following cell-depleting therapies, including investigational agents or approved therapies: CAMPATH, anti-CD4, anti-CD5, and anti-CD3.
12. Previous treatment with ABT.
13. History of severe allergic or anaphylactic reactions to monoclonal antibodies.
14. Evidence of serious uncontrolled concomitant cardiovascular, nervous system, renal, hepatic, endocrine (include uncontrolled diabetes mellitus) or gastrointestinal disease (including complicated diverticulitis, ulcerative colitis, or Crohn's disease.)
15. Evidence of concomitant lung disease which PI feels may interfere with clinical assessment of ILD for example severe active chronic obstructive pulmonary disease (COPD), asthma, occupational lung disease, pulmonary sarcoidosis, etc.
16. Prisoners or subjects who are compulsory detained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2023-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Aggarwal, MD, Principal Investigator — University of Pittsburgh
Locations (5):
- United States (5):
  - Cedars-Sinai Medical Center, Beverly Hills, California
  - University of Colorado Anschutz Medical Campus, Denver, Colorado
  - John Hopkins Medical Center, Baltimore, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurasawa K, Nawata Y, Takabayashi K, Kumano K, Kita Y, Takiguchi Y, Kuriyama T, Sueishi M, Saito Y, Iwamoto I. Activation of pulmonary T cells in corticosteroid-resistant and -sensitive interstitial pneumonitis in dermatomyositis/polymyositis. Clin Exp Immunol. 2002 Sep;129(3):541-8. doi: 10.1046/j.1365-2249.2002.01933.x. PMID 12197897
- [Background] Israel-Assayag E, Fournier M, Cormier Y. Blockade of T cell costimulation by CTLA4-Ig inhibits lung inflammation in murine hypersensitivity pneumonitis. J Immunol. 1999 Dec 15;163(12):6794-9. PMID 10586079
- [Background] Jimenez-Alvarez L, Arreola JL, Ramirez-Martinez G, Ortiz-Quintero B, Gaxiola M, Reynoso-Robles R, Avila-Moreno F, Urrea F, Pardo A, Selman M, Zuniga J. The effect of CTLA-4Ig, a CD28/B7 antagonist, on the lung inflammation and T cell subset profile during murine hypersensitivity pneumonitis. Exp Mol Pathol. 2011 Dec;91(3):718-22. doi: 10.1016/j.yexmp.2011.09.010. Epub 2011 Sep 14. PMID 21945736
- [Background] Murata K, Dalakas MC. Expression of the costimulatory molecule BB-1, the ligands CTLA-4 and CD28, and their mRNA in inflammatory myopathies. Am J Pathol. 1999 Aug;155(2):453-60. doi: 10.1016/s0002-9440(10)65141-3. PMID 10433938
- [Background] Nagaraju K, Raben N, Villalba ML, Danning C, Loeffler LA, Lee E, Tresser N, Abati A, Fetsch P, Plotz PH. Costimulatory markers in muscle of patients with idiopathic inflammatory myopathies and in cultured muscle cells. Clin Immunol. 1999 Aug;92(2):161-9. doi: 10.1006/clim.1999.4743. PMID 10444360
- [Background] Cutolo M, Soldano S, Montagna P, Sulli A, Seriolo B, Villaggio B, Triolo P, Clerico P, Felli L, Brizzolara R. CTLA4-Ig interacts with cultured synovial macrophages from rheumatoid arthritis patients and downregulates cytokine production. Arthritis Res Ther. 2009;11(6):R176. doi: 10.1186/ar2865. Epub 2009 Nov 23. PMID 19930661
- [Background] Buch MH, Boyle DL, Rosengren S, Saleem B, Reece RJ, Rhodes LA, Radjenovic A, English A, Tang H, Vratsanos G, O'Connor P, Firestein GS, Emery P. Mode of action of abatacept in rheumatoid arthritis patients having failed tumour necrosis factor blockade: a histological, gene expression and dynamic magnetic resonance imaging pilot study. Ann Rheum Dis. 2009 Jul;68(7):1220-7. doi: 10.1136/ard.2008.091876. Epub 2008 Sep 4. PMID 18772191
- [Background] Lumsden JM, Roberts JM, Harris NL, Peach RJ, Ronchese F. Differential requirement for CD80 and CD80/CD86-dependent costimulation in the lung immune response to an influenza virus infection. J Immunol. 2000 Jan 1;164(1):79-85. doi: 10.4049/jimmunol.164.1.79. PMID 10604996
- [Background] Platt AM, Gibson VB, Patakas A, Benson RA, Nadler SG, Brewer JM, McInnes IB, Garside P. Abatacept limits breach of self-tolerance in a murine model of arthritis via effects on the generation of T follicular helper cells. J Immunol. 2010 Aug 1;185(3):1558-67. doi: 10.4049/jimmunol.1001311. Epub 2010 Jul 2. PMID 20601593
- [Background] Mitsui T, Kuroda Y, Ueno S, Kaji R. The effects of FK506 on refractory inflammatory myopathies. Acta Neurol Belg. 2011 Sep;111(3):188-94. PMID 22141281
- [Background] Ochi S, Nanki T, Takada K, Suzuki F, Komano Y, Kubota T, Miyasaka N. Favorable outcomes with tacrolimus in two patients with refractory interstitial lung disease associated with polymyositis/dermatomyositis. Clin Exp Rheumatol. 2005 Sep-Oct;23(5):707-10. PMID 16173253
- [Background] Ando M, Miyazaki E, Yamasue M, Sadamura Y, Ishii T, Takenaka R, Ito T, Nureki S, Kumamoto T. Successful treatment with tacrolimus of progressive interstitial pneumonia associated with amyopathic dermatomyositis refractory to cyclosporine. Clin Rheumatol. 2010 Apr;29(4):443-5. doi: 10.1007/s10067-009-1358-x. Epub 2010 Feb 4. PMID 20130943
- [Background] Takada K, Nagasaka K, Miyasaka N. Polymyositis/dermatomyositis and interstitial lung disease: a new therapeutic approach with T-cell-specific immunosuppressants. Autoimmunity. 2005 Aug;38(5):383-92. doi: 10.1080/08916930500124023. PMID 16227154
- [Background] Wilkes MR, Sereika SM, Fertig N, Lucas MR, Oddis CV. Treatment of antisynthetase-associated interstitial lung disease with tacrolimus. Arthritis Rheum. 2005 Aug;52(8):2439-46. doi: 10.1002/art.21240. PMID 16052580
- [Background] Guglielmo S, Bertinaria M, Rolando B, Crosetti M, Fruttero R, Yardley V, Croft SL, Gasco A. A new series of amodiaquine analogues modified in the basic side chain with in vitro antileishmanial and antiplasmodial activity. Eur J Med Chem. 2009 Dec;44(12):5071-9. doi: 10.1016/j.ejmech.2009.09.012. Epub 2009 Sep 15. PMID 19811859
- [Background] Kerola AM, Nieminen TV, Kauppi MJ, Kautiainen H, Puolakka K, Virta LJ, Kerola T. Increased risk of levothyroxine-treated hypothyroidism preceding the diagnosis of rheumatoid arthritis: a nationwide registry study. Clin Exp Rheumatol. 2014 Jul-Aug;32(4):455-9. Epub 2014 Jun 6. PMID 24959977
- [Background] Arabshahi B, Silverman RA, Jones OY, Rider LG. Abatacept and sodium thiosulfate for treatment of recalcitrant juvenile dermatomyositis complicated by ulceration and calcinosis. J Pediatr. 2012 Mar;160(3):520-2. doi: 10.1016/j.jpeds.2011.11.057. Epub 2012 Jan 13. PMID 22244459
- [Background] Maeshima K, Kiyonaga Y, Imada C, Iwakura M, Hamasaki H, Haranaka M, Ishii K. Successful treatment of refractory anti-signal recognition particle myopathy using abatacept. Rheumatology (Oxford). 2014 Feb;53(2):379-80. doi: 10.1093/rheumatology/ket251. Epub 2013 Aug 6. No abstract available. PMID 23920268
- [Background] Elhai M, Meunier M, Matucci-Cerinic M, Maurer B, Riemekasten G, Leturcq T, Pellerito R, Von Muhlen CA, Vacca A, Airo P, Bartoli F, Fiori G, Bokarewa M, Riccieri V, Becker M, Avouac J, Muller-Ladner U, Distler O, Allanore Y; EUSTAR (EULAR Scleroderma Trials and Research group). Outcomes of patients with systemic sclerosis-associated polyarthritis and myopathy treated with tocilizumab or abatacept: a EUSTAR observational study. Ann Rheum Dis. 2013 Jul;72(7):1217-20. doi: 10.1136/annrheumdis-2012-202657. Epub 2012 Dec 19. PMID 23253926
- [Background] Mera-Varela A, Perez-Pampin E. Abatacept therapy in rheumatoid arthritis with interstitial lung disease. J Clin Rheumatol. 2014 Dec;20(8):445-6. doi: 10.1097/RHU.0000000000000084. No abstract available. PMID 25417684
- [Background] Khanna D, Mittoo S, Aggarwal R, Proudman SM, Dalbeth N, Matteson EL, Brown K, Flaherty K, Wells AU, Seibold JR, Strand V. Connective Tissue Disease-associated Interstitial Lung Diseases (CTD-ILD) - Report from OMERACT CTD-ILD Working Group. J Rheumatol. 2015 Nov;42(11):2168-71. doi: 10.3899/jrheum.141182. Epub 2015 Mar 1. PMID 25729034
- [Derived] Aggarwal R, Pongtarakulpanit N, Sullivan DI, Moghadam-Kia S, Bae SS, Wilkerson J, Saygin D, Marder G, Venuturupalli S, Dellaripa PF, Danoff SK, Doyle T, Hunninghake GM, Lee JS, Fischer A, Falk J, Johnson C, Koontz D, Ascherman DP, Oddis CV. Abatacept for the treatment of myositis-associated interstitial lung disease. Rheumatology (Oxford). 2025 Dec 1;64(SI):SI156-SI168. doi: 10.1093/rheumatology/keaf218. PMID 40272902
- [Derived] Bae SS, Abtin F, Kim G, Markovic D, Chan C, Moghadam-Kia S, Oddis CV, Sullivan D, Marder G, Venuturupalli S, Dellaripa PF, Doyle TJ, Hunninghake GM, Falk J, Charles-Schoeman C, Tashkin DP, Goldin J, Aggarwal R. Relationship between high-resolution computed tomography quantitative imaging analysis and physiological and clinical features in antisynthetase syndrome-related interstitial lung disease. RMD Open. 2024 Nov 27;10(4):e004592. doi: 10.1136/rmdopen-2024-004592. PMID 39608864
- [Derived] Bae SS, Markovic D, Saygin D, Sullivan D, Yamaguchi K, Moghadam-Kia S, Oddis CV, Abtin F, Kim GHJ, Marder G, Venuturupalli S, Dellaripa PF, Danoff S, Doyle T, Hunninghake G, Lee JS, Falk J, Johnson C, Goldin J, Tashkin D, Charles-Schoeman C, Aggarwal R. Associations between 6-minute walk distance and physiologic measures and clinical outcomes in myositis-associated interstitial lung disease. Rheumatology (Oxford). 2025 Dec 1;64(SI):SI79-SI87. doi: 10.1093/rheumatology/keae477. PMID 39222437

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from four clinical sites between June 2017 through May 2021.
Groups:
- Placebo: Subcutaneous placebo injection weekly for 24 weeks. 24 week optional follow up phase all subjects receive abatacept 125 mg weekly.
  Placebo: Placebo
Period: Randomized, Placebo-controlled
Arm/Group | Placebo | Abatacept
Started | 11 | 9
Completed | 11 | 8
Not Completed | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Period: Open Label Extension
Arm/Group | Placebo | Abatacept
Started | 11 | 8
Completed | 9 | 7
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Abatacept | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.95 (6.87) | 51.56 (10.69) | 53.98 (8.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 9 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 10 | 7 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Forced Vital Capacity (FVC) % [Median (Inter-Quartile Range); unit: %] | 61.0 [53.0 to 80.0] | 66.0 [49.0 to 68.5] | 63.5 [52.3 to 72.5]

OUTCOME MEASURES:

1. Primary Outcome: % Predicted Forced Vital Capacity (FVC) Absolute Change
Description: The primary outcome criteria for efficacy will be the absolute change of % predicted FVC from the baseline visit to week 24 between the 2 treatment arms (SOC/placebo vs. SOC/Abatacept).
Time Frame: 24 Weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: % predicted FVC
Arm/Group | Placebo | Abatacept
Number analyzed (Participants) | 11 | 9
% predicted FVC | -1.70 [-5.90 to 2.50] | -2.05 [-6.97 to 2.87]
Statistical Analysis 1: Comparison: Placebo vs Abatacept; The null hypothesis for the change outcomes is µABT - µPlacebo = 0; Test type: Superiority; p < 0.05, Mixed Models Analysis; Adjustments are for baseline FVC, age, and gender, with a repeated measures effect of participant; Median Difference (Net) = -2.55, 95% CI 2-sided [-9.36 to 4.26], Standard Error of Mean 3.34 — The comparison difference value is µABT - µPlacebo

2. Secondary Outcome: Time to Progression Free Survival
Description: The first occurrence of any of the following: death or lung transplantation or decline in % predicted FVC ≥ 10% or decline in % predicted FVC ≥ 5% with a decline in % predicted DLCO ≥ 15%
Time Frame: 48 weeks
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Placebo | Abatacept
Number analyzed (Participants) | 11 | 9
Weeks | 27.71 [12.71 to 46.86] | 16.86 [15.36 to 34.93]
Statistical Analysis 1: Comparison: Placebo vs Abatacept; The null hypothesis for the time to event outcomes is exp(bABT) / exp(bPlacebo) = 1; Test type: Superiority; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 0.66, 95% CI 2-sided [0.16 to 2.77], Standard Error of Mean 0.73 — ABT is the numerator and Placebo is the denominator for the hazard ratios. The dispersion value given is the SE of the estimate on the natural log scale

3. Secondary Outcome: Comparison of Change in Patient Reported Dyspnea Scores (University of California San Diego Shortness of Breath Questionnaire)
Description: Measured by University of California San Diego Shortness of Breath Questionnaire (UCSD SOBQ) (range 0-120, higher score is worsening dyspnea).
Time Frame: 24 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Placebo | Abatacept
Number analyzed (Participants) | 11 | 9
score on a scale | -4.59 [-15.54 to 6.36] | 3.20 [-8.86 to 15.26]
Statistical Analysis 1: Comparison: Placebo vs Abatacept; The null hypothesis for the change outcomes is µABT - µPlacebo = 0; Test type: Superiority; p < 0.05, Mixed Models Analysis; Adjustments are for baseline FVC, age, and gender, with a repeated measures effect of participant; Mean Difference (Net) = 7.51, 95% CI 2-sided [-8.80 to 23.83], Standard Error of Mean 8.12 — The comparison difference value is µABT - µPlacebo

4. Secondary Outcome: Time to Improvement in % Predicted FVC ≥10%
Description: Comparison of percent predicted FVC results from pulmonary function tests from baseline to week 48. Improvement is defined as a % predicted FVC change ≥10%
Time Frame: 48 weeks
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Placebo | Abatacept
Number analyzed (Participants) | 11 | 9
weeks | 17.86 [9.86 to 25.86] | 11.86 [11.86 to 11.86]
Statistical Analysis 1: Comparison: Placebo vs Abatacept; The null hypothesis for the time to event outcomes is exp(bABT) / exp(bPlacebo) = 1; Test type: Superiority; p < 0.05, Regression, Cox; Hazard Ratio (HR) = 0.42, 95% CI 2-sided [0.04 to 4.02], Standard Error of Mean 1.16 — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Baseline (week 0) through end of study Visit 5 (week 48)
Arm/Group | Placebo | Abatacept
All-Cause Mortality (participants affected / at risk) | 0/11 | 1/20
Serious Adverse Events (participants affected / at risk) | 0/11 | 3/20
Other Adverse Events (participants affected / at risk) | 5/11 | 6/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=11) | Abatacept (N=20)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Unrelated serious adverse event that resulted in death due to worsening disease
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Placebo (N=11) | Abatacept (N=20)
Excessive bruising (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Eye Infection (Infections and infestations) | 0 (0) | 1/9 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Infection (Infections and infestations) | 2 (2) | 3 (3)
Lip infection (Infections and infestations) | 0 (0) | 1 (1)
Deceased lymphocyte count (Investigations) | 0 (0) | 2 (2)
Aspartate aminotransferase (Investigations) | 1 (1) | 0 (0)
alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Decreased DLCO (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1)
Oral thrush (Infections and infestations) | 0 (0) | 1 (1)
Chest pain (Cardiac disorders) | 0 (0) | 2 (2)
colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (3)
oral mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
pain in extremities (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
renal calculi (Renal and urinary disorders) | 0 (0) | 2 (2)
voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
other (Reproductive system and breast disorders) | 0 (0) | 1 (1)
dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
rash on extremities (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/27/NCT03215927/Prot_SAP_002.pdf
  • Informed Consent Form (2019-01-23): https://cdn.clinicaltrials.gov/large-docs/27/NCT03215927/ICF_003.pdf